CLINICAL TRIAL: NCT04873232
Title: A 6-Month Extension Study Following Protocol VMDN-003-2 - An Adaptive, Phase 3, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess Engensis in Participants With Painful Diabetic Peripheral Neuropathy
Brief Title: A 6-Month Extension Study of VMDN-003-2 to Assess Engensis in Participants With Painful Diabetic Peripheral Neuropathy
Acronym: REGAiN-1B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMDN-003-2b
Record Dates: First submitted 2021-02-18; First posted 2021-05-05 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Engensis (Experimental): Patients who have received Engensis in protocol VMDN-003-2
  Interventions: Biological: Engensis
- Placebo (Placebo Comparator): Patients who have received Placebo in protocol VMDN-003-2
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Engensis — Injections with Engensis in study VMDN-003-2
  Arms: Engensis
Other: Placebo — Injections with Placebo in study VMDN-003-2
  Arms: Placebo

SUMMARY:
To evaluate the durability of efficacy and long-term safety of intramuscular administration of Engensis or Placebo that was administered in the double-blind, randomized, VMDN-003-2 Placebo-controlled Phase 3 Study.

DETAILED DESCRIPTION:
The purpose of this 6-month extension study (VMDN-003-2b) is to evaluate the durability of efficacy and long-term safety of intramuscular administration of Engensis or Placebo that was administered in the double-blind, randomized, VMDN-003-2 Placebo-controlled Phase 3 Study. No treatments will be administered in this VMDN-003-2b extension study. The combined overall duration of the VMDN-003-2 and VMDN-003-2b studies will be 12 months.

Participants will be enrolled in the VMDN-003-2b study at completion of the Day 180 Visit of Study VMDN-003-2. Participants will continue to be identified by the same Participant number and the same treatment group (Engensis or Placebo) assigned by randomization in Study VMDN-003-2. No study drug or treatment will be administered in this VMDN-003-2b extension study. The double-blind treatment assignment from the prior study will be maintained for Investigators and Participants during this extension study.

This extension study will assess the durability of efficacy and long-term safety of Engensis compared to Placebo as measured by changes in Average Daily Pain Score of the full Brief Pain Inventory for Diabetic Peripheral Neuropathy, Bedside sensory testing, physical examinations, laboratory assessments, vital signs, treatment-emergent adverse events, treatment-emergent serious adverse events, and adverse events of special interest.

ELIGIBILITY:
Inclusion Criteria:

* Completed study VMDN-003-2 and consent to enroll in study VMDN-003-2b

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2024-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Arizona Research Center, Phoenix, Arizona
  - Clinical Trials - Little Rock, Little Rock, Arkansas
  - California Medical Clinic for Headache, Los Angeles, California
  - Clinical Trials Research - Sacramento, Sacramento, California
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Gateway Clinical Trials, LLC, O'Fallon, Illinois
  - Foot & Ankle Center of Illinois, Springfield, Illinois
  - Clinical Research Professionals, Chesterfield, Missouri
  - Richmond Behavioral Associates, Staten Island, New York
  - Health Concepts, Rapid City, South Dakota
  - Nerve and Muscle Center of Texas, Houston, Texas
  - Futuro Clinical Trials, McAllen, Texas
  - ClinPoint Trials LLC, Waxahachie, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Dominion Medical Associates, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Qualified subjects were anyone that completed the Day 180 visit in VMDN-003-2 (NCT04469270) and provided informed consent to be followed for another 6 months in this extension protocol VMDN-003-2b (NCT04873232). Subjects did not receive any further investigational prouct interventions.
Period: Overall Study
Arm/Group | Engensis | Placebo
Started | 49 | 57
Completed | 47 | 53
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engensis | Placebo | Total
Number analyzed (Participants) | 49 | 57 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 34 | 63
  >=65 years | 20 | 23 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 31 | 43 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 42 | 49 | 91
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 17 | 26
  White | 37 | 36 | 73
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Efficacy of Intramuscular Administration of Engensis on Reducing Pain in Participants With Painful Diabetic Peripheral Neuropathy in the Feet and Lower Legs as Compared to Placebo
Description: Change in the means of the Average Daily Pain Scores from the full Brief Pain Inventory for Diabetic Peripheral Neuropathy from the 7 days prior to the Day 0 Visit (Study VMDN-003-2) to the 7 days prior to the Day 365 Visit in the intent-to-treat population. The mean of the Average Daily Pain Scores are used for the primary endpoint recorded in the 7 days prior to the Days 270 and 365/ET Visits. The Brief Pain Inventory for Diabetic Peripheral Neuropathy scale is a 0 to 10 point scale with 10 being Pain as bad as you can imagine.
  The mean of at least 5 daily pain scores recorded for Question 5 of the Brief Pain Inventory for Diabetic Peripheral Neuropathy scale in electronic diary during the 7 days prior to the visits on Days 270 and 365/Early termination. The greater the negative difference between the followup visit and the Day 0 Baseline for each group for the average daily pain score in participants, would indicate that the average daily pain is declining.
Time Frame: From the 7 days prior to the Day 0 Visit (Study VMDN-003-2, NCT04469270), Day 270, to the 7 days prior to the Day 365 Visit in the intent-to-treat population
Population: Summary of Change from Baseline to Day 365 in ADPS (Intent-To-Treat Population)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 49 | 57
score on a scale
  Change from Baseline to Day 270: number analyzed (Participants) | 47 | 52
  Change from Baseline to Day 270 | -2.27 (2.083) | -2.62 (2.087)
  Change from Baseline to 7 Days prior to the Day 365 visit: number analyzed (Participants) | 43 | 49
  Change from Baseline to 7 Days prior to the Day 365 visit | -2.53 (2.173) | -2.78 (2.126)

2. Secondary Outcome: To Evaluate the Efficacy of IM Administration of Engensis on the Worst Pain in Participants With Painful Diabetic Peripheral Neuropathy in the Feet and Lower Legs as Compared to Placebo
Description: Change in the means of the Worst Pain Scores from the full Brief Pain Inventory for Diabetic Peripheral Neuropathy from the 7 days prior to Day 0 Visit (Study VMDN-003-2), to Day 270, and 7 days prior to the Day 365 Visit for Engensis compared to Placebo. The Brief Pain Inventory for Diabetic Peripheral Neuropathy scale is a 0 to 10 point scale with 10 being Pain as bad as you can imagine.
  The mean of at least 5 worst daily pain scores recorded for Question 3 of the Brief Pain Inventory for Diabetic Peripheral Neuropathy in the electronic diary during the 7 days prior to the Visits on Days 270 and 365/Early termination. The greater the negative difference between the followup visit and the Day 0 Baseline for each group for the worst pain score in participants, would indicate that the worst pain is declining.
Time Frame: From the 7 days prior to the Day 0 Visit (Study VMDN-003-2) to the 7 days prior to the Day 365 Visit for Engensis compared to Placebo
Population: Summary of Change from Day 0, Baseline, to Day 270, and Day 365 in Worst Pain Score (MI) (Intent-To-Treat Population)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 49 | 57
units on a scale
  Change from Baseline to Day 270: number analyzed (Participants) | 47 | 52
  Change from Baseline to Day 270 | -2.50 (2.376) | -2.94 (2.664)
  Change from Baseline to Day 365: number analyzed (Participants) | 43 | 49
  Change from Baseline to Day 365 | -2.65 (2.485) | -3.19 (2.454)

3. Secondary Outcome: To Evaluate the Safety of IM Administration of Engensis in the Number of Participants With Painful DPN in the Feet and Lower Legs as Compared to Placebo
Description: Number of participants with adverse events and serious adverse events for Engensis compared to Placebo, including the number of participants with clinically significant laboratory values for Engensis compared to Placebo
Time Frame: From Day 0 Visit (Study VMDN-003-2) to the Day 365 Visit
Population: Overall Summary of number of participants with Adverse Events (Safety Population)
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 49 | 57
Participants | 16 | 22

4. Secondary Outcome: To Evaluate the Efficacy of Administration of Engensis on Reducing Pain in Participants With Painful Diabetic Peripheral Neuropathy in the Feet and Lower Legs
Description: Proportion of Responders (≥ 50% reduction in the Average Daily Pain Scores from the full Brief Pain Inventory for Diabetic Peripheral Neuropathy) from the 7 days prior to the Day 0 Visit (Study VMDN-003-2) to the 7 days prior to the Day 270 Visit and the 7 days prior to the Day 365 Visit for Engensis compared to Placebo.
Time Frame: From the 7 days prior to the Day 0 Visit (Study VMDN-003-2), to the 7 days prior to the Day 270 Visit, and 7 days prior to the Day 365 Visit
Population: Summary of Participant Responders with ≥50% reduction from Baseline Day 0 visit, in the Average Daily Pain Score to the 7 days prior to Day 270 and 7 days prior to the Day 365 visit (Intent-To-Treat Population)
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 49 | 57
Participants
  Responders with ≥50% reduction by Day 270 | 17 | 27
  Responders with ≥50% reduction by Day 365 | 16 | 27

ADVERSE EVENTS:
Time Frame: Adverse events that started after the Day 180 Visit (Day 180 Visit date +1 day), and recorded up to the end of the study visit, Day 365.
Description: For each category, participants were included only once, even if they experienced multiple events in that category. Treatment-emergence was defined as adverse events that occurred the day after Day 180 Visit (Day 180 Visit date +1 day), and recorded by the end of the study visit, Day 365.
  Two participants signed informed consent but never returned for follow-up visits so Adverse Event information for them could not be collected.
Arm/Group | Engensis | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/57
Serious Adverse Events (participants affected / at risk) | 3/49 | 6/57
Other Adverse Events (participants affected / at risk) | 16/49 | 22/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engensis (N=49) | Placebo (N=57)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engensis (N=49) | Placebo (N=57)
COVID-19 (Infections and infestations) | 2 (2) | 3 (3)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Gastoenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 1 (1)
Conjunctival oedema (Eye disorders) | 0 (0) | 1 (1)
Dry age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine abnormal (Investigations) | 0 (0) | 1 (1)
Blood urea abnormal (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is NOT an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT04873232/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/32/NCT04873232/SAP_001.pdf